CLINICAL TRIAL: NCT04194099
Title: Development and Application of a Novel Neurorehabilitation Technology With Paired Associative Nerve Stimulation in Spinal Cord Injured Subjects
Brief Title: Effects of Paired Associative Nerve Stimulation on Spinal Cord Injury Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Lai chien hung, Professor, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201905031
Record Dates: First submitted 2019-12-05; First posted 2019-12-11 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Trans-cranial magnetic stimulation; Trans-spinal direct current stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- rTMS (Brain) + tsES (Spinal) (Experimental): First part 20 Hz rTMS (Brain) + Anode tsDCS (Spinal)
  Brain:
  1. Train pulse: 2 sec
  2. Inter-train: 28 sec
  3. Total time: 1200 sec
  Spinal:
  Continuous direct current (DC): 1200 sec
  Second part iTBS rTMS(Brain) + 2.5-mA tsDCS (Spinal)
  Brain:
  1. Train pulse: 2 sec
  2. Inter-train: 8 sec
  3. Total time: 200 sec
  Spinal:
  Continuous direct current (DC): 600 sec
  Interventions: Device: 20 Hz rTMS (Brain); Device: Anode tsDCS (Spinal)
- rTMS (Brain) + tsES (Spinal) or sham stimulation (Experimental): First part 20 Hz rTMS (Brain) + 20 Hz current square-wave pulses (Spinal)
  Brain and spinal:
  1. Train pulse: 2 sec
  2. Inter-train: 28 sec
  3. Total time: 1200 sec
  Second part iTBS rTMS(Brain) + sham 2.5-mA tsDCS (Spinal)
  Brain:
  1. Train pulse: 2 sec
  2. Inter-train: 8 sec
  3. Total time: 200 sec
  Spinal:
  Sham direct current (DC) stimulation
  Interventions: Device: 20 Hz rTMS (Brain); Device: 20 Hz current square-wave pulses (Spinal)
- iTBS rTMS or sham (Brain) + tsES or sham (Spinal) (Experimental): First part
  Brain:
  1. Train pulse: 2 sec
  2. Inter-train: 8 sec
  3. Total time: 200 sec
  Spinal:
  Continuous direct current (DC): 190 sec
  Second part Sham iTBS rTMS (Brain) + 2.5-mA tsDCS (Spinal)
  Sham iTBS rTMS Brain:
  Spinal:
  Continuous direct current (DC): 600 sec
  Interventions: Device: iTBS rTMS (Brain); Device: Anode tsDCS (Spinal)
- iTBS rTMS or sham (Brain) + iTBS or sham (Spinal) (Experimental): First part
  Brain and spinal:
  1. Train pulse: 2 sec
  2. Inter-train: 8 sec
  3. Total time: 200 sec
  Second part Sham iTBS rTMS (Brain) + Sham 2.5-mA tsDCS (Spinal)
  Brain:
  Sham iTBS rTMS
  Spinal:
  Sham direct current (DC) stimulation
  Interventions: Device: iTBS rTMS (Brain); Device: iTBS (Spinal)
- sham (no stimulation on brain nor spinal) (Sham Comparator): First part Sham stimulation.
  No second part
  Interventions: Device: sham

INTERVENTIONS:
Device: 20 Hz rTMS (Brain) — Higher frequency (>5 Hz) trains increase cortical excitability.
  Arms: rTMS (Brain) + tsES (Spinal); rTMS (Brain) + tsES (Spinal) or sham stimulation
Device: iTBS rTMS (Brain) — Intermittent theta burst stimulation (iTBS) is a newer rTMS approach.
  Arms: iTBS rTMS or sham (Brain) + iTBS or sham (Spinal); iTBS rTMS or sham (Brain) + tsES or sham (Spinal)
Device: Anode tsDCS (Spinal) — Anodal tsDCS increased the spinal reflex amplitude, as well as corticospinal excitability.
  Arms: iTBS rTMS or sham (Brain) + tsES or sham (Spinal); rTMS (Brain) + tsES (Spinal)
Device: 20 Hz current square-wave pulses (Spinal) — Higher frequency (>5 Hz) of current increase cortical excitability.
  Arms: rTMS (Brain) + tsES (Spinal) or sham stimulation
Device: iTBS (Spinal) — Intermittent theta-burst stimulation (iTBS) is a newer approach. it may increase corticospinal excitability.
  Arms: iTBS rTMS or sham (Brain) + iTBS or sham (Spinal)
Device: sham — with sham stimulation on brain and spinal.
  Arms: sham (no stimulation on brain nor spinal)

SUMMARY:
This study is to investigate the effects of repetitive transcranial magnetic stimulation (rTMS) combined with trans-spinal electrical stimulation (tsES) intervention on cortical excitability, brain structure, motor ability of lower limb in individuals with incomplete spinal cord injury. Twelve participants will be recruited in this study.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) impairs motor and sensory function and affects numerous body functions and daily activities. Insufficient central nervous system plasticity can result in maladaptive changes that prevent full recovery. It's a challenge to guide this plasticity to optimize the functional outcome for individuals with SCI.

Transcranial magnetic stimulation (TMS) and trans-spinal electric stimulation (tsES) may modulate cortical excitability, corticospinal output and spinal circuit. However, few studies investigated the effectiveness of paired nerve stimulation (PNS) on neuroplasticity and functional outcome in persons with SCI. Therefore, this study aim to examine the effects of the combination of these two different non-invasive nerve stimulation with the cycling exercise on the motor cortex and corticospinal circuit excitability as well as functional recovery.

Present study clarifies the effects of five different settings of combined with TMS and tsES intervention and then undergo cycling exercise after PNS on spinal cord and cortical excitability in SCI participants.

It is expected that this project will successfully establish a new neuromodulation technology to enhance cortical, corticospinal and spinal circuit excitability as well as to improve the outcome of lower-limb function and quality of life in persons with SCI. Therefore, this project can not only publish scientific papers, but also can enhance the neuroplasticity and improve function in persons with SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 to 65 years incomplete SCI (American Spinal Injury Association Impairment Scale (ASIA) B to D)
2. Lesion area above the tenth thoracic vertebra (T10)
3. Injury time more than one year
4. Without range of motion (ROM) limitation
5. Medical condition stable

Exclusion Criteria:

1. Having pacemaker, cochlear implants, metal in the brain or skull, open wound of brain, or history of epilepsy.
2. Having seizure history
3. Having other neurological, mental, medical problems affect this study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Motor evoked potentials (MEP) | Just before the intervention start and immediately after the intervention finished.
  Motor evoked potential (MEP) is recorded from tibialis anterior muscles following direct transcranial magnetic stimulation (TMS) of motor cortex. All TMS is delivered with the participant seated upright on the chair. Both passive and active conditions, participants are instructed to relax their one hand in the seated position. TMS is delivered over the motor cortex (M1) using a concave double cone coil (Magstim Co., United Kingdom) attached to a BiStim magnetic stimulator (Magstim Co., United Kingdom). To locate the optimized site, stimuli are delivered over various points around the Cz (approximate 1 cm distance from Cz). The optimal site is the location around the Cz that evoked the greatest MEP amplitude in tibialis anterior muscles. The onset latency and onset to peak amplitude will be assessed.
Change of resting motor threshold (RMT) | Just before the intervention start and immediately after the intervention finished.
  Resting motor threshold (RMT) is recorded from tibialis anterior muscles following transcranial magnetic stimulation. TMS is delivered over the motor cortex (M1) using a concave double cone coil (Magstim Co., United Kingdom) attached to a BiStim magnetic stimulator (Magstim Co., United Kingdom). To locate the optimal site, stimuli are delivered over various points around the Cz (the distance approximate 1 cm from Cz) to get the hot spot point. And then measure the RMT using the minimum stimulus intensity that produced a minimal motor evoked response (about 50 micro-volts (µV) in at least 5 of 10 trials) at rest.

SECONDARY OUTCOMES:
Change of Modified Ashworth Scale (MAS) | Just before the intervention start and immediately after the intervention finished.
  Modified Ashworth scale (MAS) measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. Scoring is recorded as follows:
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the Range of motion (ROM)
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
Change of Lower Extremities Motor Score (LEMS) | Just before the intervention start and immediately after the intervention finished.
  The voluntary muscle strength of five key muscles (hip flexors, knee extensors, ankle dorsiflexors, long toe extensors and ankle plantarflexors) of both lower extremities was tested.
  Each muscle was given a value between 0 and 5 according to the strength of voluntary muscle contraction.
  Maximum and minimum LEMS were 50 and 0, respectively.
Change of functional Magnetic Resonance Imaging (fMRI) | Immediately after the intervention finished.
  Our study will use 3 Tesla (T) magnetic resonance imaging[GE DISCOVERY MR750w system (GE Healthcare, Milwaukee, Wisconsin)] for functional magnetic resonance imaging. Resting-state functional MRI image is an echo-planar Image (EPI) technique, using a parameter time of repetition of 2500 milliseconds, time of echo is 30 milliseconds, 43 axial slices, slice thickness is 3 mm, flip angle is 80 degrees, field of view is 192 × 192 mm, and vixen size is 3 × 3 × 3 mm. The EPI scan for 525 seconds. All subjects are asked to close their eyes and supine. Our study uses the fractional amplitude of low-frequency fluctuations analysis to confirm abnormal brain function.
Change of Surface Electromyography (sEMG) | Just before the intervention start and immediately after the intervention finished.
  sEMG recordings using pairs of 1 cm-diameter silver/silver chloride recessed sEMG electrodes placed over the muscle bellies 3 cm apart were made from the right and left quadriceps (mainly rectus femoris) and hamstrings.
  Electrodes were centered on the long axis over muscle bellies for recording during voluntary motor tasks performed by 30 min cycling exercise.
  The 4 sEMG channels were recorded with a bandwidth of 30 to 500 Hz and a gain of 1,000. Movement sensor and event cue marker outputs were also recorded and, along with the sEMG, were continually digitized at a rate of 2,000 samples/s for the duration of the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Lai, MD PhD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical university Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No